CLINICAL TRIAL: NCT02343887
Title: CogStim, a Pilot Study : Cognitive Rehabilitation Management of HIV-1 Mild Cognitively Impaired Patients Controlled With Antiretroviral Therapy
Acronym: CogStim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013-49; 2013-A01621-44 (Other: ansm)
Record Dates: First submitted 2014-11-14; First posted 2015-01-22 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: HIV
MeSH Terms: interventions — Neuropsychological Tests; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (Active Comparator): patients without taking into cognitive or psychological treatment for 6 months (period 1) and
  * if the situation improves in the neuropsychological assessment of M6 further with simple monitoring neuropsychological evaluation M12
  * or persistence or worsening of the disorder, the beginning of a cognitive remediation program for 6 months (period 2).
  Interventions: Other: neuropsychological tests; Other: STAI-Y scale for anxiety; Other: Beck scale for depression; Other: without intervention
- group with cognitive rehabilitation, (Experimental): patients treated for 6 months Cognitive remediation (period 1), then
  * Stop if the situation improves in the evaluation and monitoring of M6 to M12 with neuropsychological assessment,
  * or persistence or worsening of the disorder, further cognitive remediation for 6 months (period 2).
  Interventions: Other: neuropsychological tests; Other: STAI-Y scale for anxiety; Other: Beck scale for depression
- group with psychological support. (Experimental): patients treated with counseling for six months (period 1) and
  * Stop if the situation improves with neuropsychological assessment and monitoring to M12,
  * or if persistent or worsening unrest in the neuropsychological assessment of M6, the beginning of a cognitive remediation program for 6 months (period 2).
  Interventions: Other: neuropsychological tests; Other: STAI-Y scale for anxiety; Other: Beck scale for depression

INTERVENTIONS:
Other: neuropsychological tests
Other: STAI-Y scale for anxiety
Other: Beck scale for depression
Other: without intervention
  Arms: control group

SUMMARY:
Despite undetectable plasma viral load under treatment, about 30% of HIV infected patients show asymptomatic neurocognitive impairment or minor cognitive disorder. These symptoms impact the compliance of the treatment, though its performance and daily life quality. To this day, no therapy tested has proved its efficiency, including the strategy of the antiretroviral therapy (cART) optimization according to the Cerebral Penetration effectiveness Score (CPE).

Description of the study: an open prospective comparative monocentric pilote study, randomised in three groups which investigates the efficiency of a 6 months-cognitive rehabilitation program on improving asymptomatic or minor cognitive disorder for undetectable HIV+ patients. This study gathers HIV-1 patients undetectable under stable cART with a good cerebral penetration who develop asymptomatic or minor cognitive disorders connected to HIV infection. Those who have severe psychiatric disorder or who are on medication that could interfere with psychometrical tests will be excluded.

Main Objective: to compare the impact of a cognitive rehabilitation program over a 6 months period on the evolution of minor cognitive disorders and asymptomatic patients to a control group and a group treated with psychological support.

DETAILED DESCRIPTION:
This is an open prospective comparative monocentric study, pilote, that randomised 60 patients in three groups of 20. This study will select 18 to 55 years old patients, with HIV infection controlled under antiretroviral therapy stble for 12 months and cognitive impairment objective on two neuropsychological evaluations separated from 6 months at least. All selected patients must have been explored by cerebral RMN or scanner

ELIGIBILITY:
Inclusion Criteria:

* - Seropositive for HIV-1 Patient
* With a plasma viral load below the limit of detection for minimum 6 months (HIV viral load <40 copies / ml)
* On stable antiretroviral therapy for 12 months, according to the revised optimized subject to the constraints of genotypic resistance and CPE score in the absence of cons-indication to treatment intensive brain penetration (Annex 15)
* With cognitive complaint objectified by the cognitive complaint questionnaire (Appendix 9: score 3 or 1 positive response among the items C4, C5, C7, C8) and cognitive impairment found by an alteration of at least two cognitive fields assessed by psychometric tests for at least 6 months
* 18 <age <55 years
* No defined by a marked depression scale score of Beck <16 (Appendix 13)
* No marked anxiety defined by a T score> 55 on the scale of Spielberger STAI-Y (Annex 14)
* Insured under the social security
* Who signed the consent form.
* Recent brain imaging excluding other causes of cognitive impairment (MRI or CT brain injected injected so-indication against MRI)

Exclusion Criteria:

* A patient diagnosed and followed for more than six months psychiatric disorder that could interfere with psychometric assessment
* Patients with a poor understanding of French,
* Patients with active opportunistic infection of the CNS or with neurological sequelae.
* History of head trauma
* Active Substance excluding cannabis
* Patient for which a change of antiretroviral therapy is provided within 12 months
* Patient for which interferon treatment is provided within 12 months
* Patient placed under guardianship,
* Patient with HIV-related dementia
* Liver cirrhosis Child B or C (Annex 16)
* Severe renal impairment (creatinine clearance by Cockcroft <30 ml / min)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
cognitive remediation strategy (BREF test) | 6 months
  - BREF test
cognitive remediation strategy (grooved pegboard test) | 6 months
  - grooved pegboard test
cognitive remediation strategy (RLRI-16 test6.) | 6 months
  - RLRI-16 test6.
cognitive remediation strategy (Digit Symbol Substitution Test) | 6 months
  - Digit Symbol Substitution Test

SECONDARY OUTCOMES:
impact on daily life quality (SF-12 Medical Outcomes Study Short-Form General Health Survey) | 6 months
  SF-12 Medical Outcomes Study Short-Form General Health Survey"
impact on daily life quality (Trail Making Test) | 6 months
  -Trail Making Test

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Paca, France